CLINICAL TRIAL: NCT05211284
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of Saroglitazar Magnesium for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD) in People Living With Human Immunodeficiency Virus (HIV) in the US
Brief Title: Saroglitazar Magnesium 4 mg for Nonalcoholic Fatty Liver Disease (NAFLD) in People Living With HIV in the US
Acronym: SARONAPLUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.20.001
Record Dates: First submitted 2022-01-24; First posted 2022-01-27 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Saroglitazar Magnesium; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar

STUDY DESIGN:
Intervention Model Description: This phase 2a study is a randomized, placebo-controlled, double-blind, parallel arm trial to evaluate the safety and efficacy of Saroglitazar Magnesium 4 mg compared with placebo in biopsy-proven NAFLD in people living with HIV (PLWH). Eligible participants will be randomized in a 1:1 ratio to receive Saroglitazar Magnesium 4 mg or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saroglitazar Magnesium 4 mg (Experimental): Saroglitazar Magnesium 4 mg tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment (24 weeks)
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Placebo Arm (Placebo Comparator): Placebo tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment (24 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar Magnesium 4 mg — Subjects randomized to Saroglitazar Magnesium 4 mg arm will receive Saroglitazar Magnesium 4 mg treatment until the duration of treatment (24 weeks).
  Arms: Saroglitazar Magnesium 4 mg
Drug: Placebo — Subjects randomized to Placebo arm will receive Placebo treatment until the duration of treatment (24 weeks).
  Arms: Placebo Arm

SUMMARY:
Saroglitazar Magnesium 4 mg for NAFLD in People Living with HIV in the US

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of Saroglitazar Magnesium for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD) in People Living with Human Immunodeficiency Virus (HIV) in the US

The four participants enrolled on version 3.0 protocol were terminated as the primary endpoint was revised from biopsy to an imaging-based approach in the subsequent protocol version 4.0. These changes were done due to recruiting challenges pertaining to biopsy. However, no participants were enrolled in the revised protocol (version 4.0) as, by then the decision to terminate the study was taken by the Sponsor considering the modifications in the internal R&D focus and a revised commercialization strategy.

The version 3.0 protocol is dated 02/Jun/2022.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age) with documented HIV.
2. Documented diagnosis of NAFLD established by imaging (ultrasound, CT scan or MRI) or liver biopsy within 6 months before screening, based on American Association for the Study of Liver Disease [AASLD] criteria
3. Hepatic fat fraction ≥8% by MRI-PDFF
4. ALT level ≥31 U/L in men and ≥19 U/L in women at Visit 1 and 2
5. HIV-1 RNA <200 copies/mL for ≥6 months on ART (must have screening HIV-1 RNA value and one clinical care value within 6 months prior to screening and up to the randomization that meets the criteria).
6. Stable ART regimen for ≥3 months prior to screening and stable up to the randomization and no active plans to change ART while on study.
7. Willingness to participate in the study.

Exclusion Criteria:

1. History of significant alcohol consumption (defined as >2 drinks/day on average for men, >1 drinks/day on average for women) for at least 3 consecutive months (12 consecutive weeks) within 5 year before screening (Note 1: 1 drink =12 ounces of beer, 8-9 ounces of malt liquor, 4 ounces of wine or 1 ounce of spirits/hard liquor. Note 2: Use sex assigned at birth for alcohol consumption limits).
2. History of other acute or chronic liver disease, including, but not limited to autoimmune, primary biliary cholangitis, Wilson's disease, alpha 1 antitrypsin deficiency, hemochromatosis, hepatitis B virus (HBV), and ongoing or recent (within the past 3 years) hepatitis C RNA positivity. (Exceptions: a. Participants with previously treated hepatitis C infection are eligible for consideration if their sustained virologic response was achieved more than 3 years prior to screening. The proportion of such participants in this trial will not exceed 25% of the study cohort. b. Participants with prior acute HBV infection that is resolved but currently do not have hepatitis B surface antigen (HBsAg) or detectable HBV DNA are eligible).
3. History of liver transplant.
4. Liver biopsy or radiologic imaging consistent with the clinical presence of cirrhosis or portal hypertension at screening.
5. Participants whose Visit 2 ALT, AST, or alkaline phosphatase (ALP) values exceed their Visit 1 values by more than 50%.

   Note: These participants will be required to have a third value measured at-least one week after V2, to assess for a trend. If the third value shows a continued increase ≥10% compared to the Visit 2 values, the participant is considered ineligible for randomization.
6. Ongoing use of steatogenic medications or supra-physiologic hormonal therapies (Exception: transgender women on stable (≥3 month) feminizing hormonal therapy not excluded), within 3 months prior to screening until time of randomization or anticipated use of medications that cause significant changes in weight during the study period (Refer Appendix 7 of protocol for 'List of Steatogenic Medications Or Supra-Physiologic Hormonal Therapies Or Medications That Cause Significant Weight Change').
7. Uncontrolled T2DM, defined as HbA1c >9.5% at screening.
8. Any of the following laboratory values at screening:

   1. ALT or AST >250 U/L
   2. Total bilirubin >1.5 mg/dL and direct bilirubin > 0.5 mg/dL (unless due to Gilbert's disease or atazanavir use per the opinion of the site investigator)
   3. Platelet count <150,000/mm3
   4. Estimated glomerular filtration rate (e-GFR) <60 mL/min/1.73m2 using the chronic kidney disease-epidemiology collaboration (CKD-EPI) equation (Refer Appendix 6 of protocol for 'CKD-EPI Calculator')
   5. International normalized ratio (INR) >1.3.
   6. Albumin < 3.6 g/dL
9. History of malignancy in the past 5 years and/or active neoplasm with the exception of superficial, non-melanoma, skin cancer.
10. Unstable cardiovascular disease, including:

    1. Unstable angina, (i.e., new or worsening symptoms of coronary heart disease) and/or acute myocardial infarction within the 3 months preceding screening
    2. Acute coronary syndrome or coronary artery intervention within the 3 months preceding screening,
    3. Heart failure of New York Heart Association (NYHA) class (III-IV) or worsening congestive heart failure within the 6 months preceding screening.
    4. History of (within 3 months preceding screening) or current unstable cardiac dysrhythmias.
    5. Uncontrolled hypertension (systolic blood pressure [SBP] >155 mmHg and/or diastolic blood pressure [DBP] >95 mmHg) at screening.
    6. Stroke or transient ischemic attack within the 6 months preceding screening.
11. Unstable pulmonary disease (based upon site investigator's evaluation) at screening.
12. Use of drugs that are known CYP2C8 inhibitors/substrates (Refer Appendix 2 of protocol for the 'List of Known CYP2C8 Inhibitors/Substrates') in the last 28 days prior to screening.
13. History of severe illness or any other conditions that require systematic treatment/or hospitalization, until participant either completes therapy or is clinically stable on therapy as per the opinion of the investigator, for at least 7 days prior to screening (such as poorly controlled psychiatric disease, active gastrointestinal conditions that might interfere with drug absorption, etc.).
14. Use of thiazolidinediones or Telmisartan within 3 months prior to screening or until time of randomization.
15. Use of unstable doses of SGLT2 inhibitors (e.g. canagliflozin, empagliflozin, dapagliflozin, etc.), glucose-dependent insulinotropic polypeptide (GIP) and/or GLP-1 agonists (e.g. semaglutide, exenatide, liraglutide, lixisenatide, tirzepatide etc.) within 6 months prior to screening until time of randomization.
16. Use of pentoxifylline, ursodeoxycholic acid, antioxidants such as vitamin E (>200 IU/day), glutathione, orlistat, betaine, or non-prescribed complementary alternative medications within 6 months prior to screening until time of randomization.
17. Known allergy, sensitivity or intolerance to the study medication or formulation ingredients.
18. History of any known bleeding disorder or coagulopathy.
19. Any condition that in the opinion of the site investigator, would compromise the participant's ability to participate in the study.
20. Unstable doses of anti-diabetic agents including sulfonylureas, biguanides or DPP-4 inhibitors in the last 3 months prior to screening until time of randomization.
21. Unstable doses of lipid lowering agents such as statins (e.g. simvastatin, pravastatin, atorvastatin, fluvastatin, lovastatin, rosuvastatin, etc.) or fibrates (clofibrate, Fenofibrate) in the last 3 months prior to screening until time of randomization.
22. Participant with weight change >5% within 6 months prior to screening until time of randomization.
23. History of bariatric surgery or currently undergoing evaluation for bariatric surgery.
24. Participation in another interventional clinical study and/or receipt of any other investigational medication within 3 months prior to screening.
25. History of COVID-19 infection in the last 30 days prior to screening.
26. Pregnancy-related exclusions, include:

    1. Pregnant/lactating female (including positive pregnancy test at screening)
    2. Pregnancy should be avoided by male and female participants either by complete abstinence or the use of acceptable effective contraceptive measures for the duration of the study and for at least 1 month after the end of the study treatment. Refer Appendix 3 Contraceptive Guidance 27. Participants having an absolute contraindication to MRI (eg., any implants, magnetic metals, cardiac pacemakers, neurostimulator) as per investigators' discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, Study Director — Zydus Therapeutics Inc.
Locations (8):
- United States (8):
  - Zydus US004, Birmingham, Alabama
  - Zydus US005, La Jolla, California
  - Zydus US006, San Francisco, California
  - Zydus US002, Indianapolis, Indiana
  - Zydus US003, Baltimore, Maryland
  - Zydus US001, Durham, North Carolina
  - Zydus US007, Houston, Texas
  - Zydus US008, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1
Not completed — Study Terminated | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Hepatic Fat Content Measured by MRI Proton Density Fat Fraction (MRI PDFF)
Description: Change from baseline in hepatic fat content
Time Frame: Week 24/EOT
Population: The 4 participants were enrolled under protocol V3.0, with biopsy-driven primary endpoint. Due to recruitment challenges, the outcome measure was modified to MRI-PDFF in the protocol V4.0. All 4 participants were prematurely terminated before completing their planned treatment before any efficacy data could be collected. No participants were enrolled under the revised protocol V4.0 as the study was terminated. Consequently, no MRI-PDFF based efficacy data were collected or analyzed
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Reduction of Hepatic Fat Content as Measured by MRI PDFF.
Description: Proportion of participants with reduction of at least 30% in hepatic fat content from baseline
Time Frame: Week 24/EOT
Population: The 4 participants were enrolled under protocol V3.0, with biopsy-driven primary endpoint. Due to recruitment challenges, the outcome measure was modified to MRI-PDFF in the protocol V4.0. All 4 participants were prematurely terminated before completing their planned treatment and before any efficacy data could be collected. No participants were enrolled under the revised protocol V4.0 as the study was terminated. Consequently, no MRI-PDFF based efficacy data were collected or analyzed
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in FibroScan®/VCTE .
Description: Change from baseline in Liver Stiffness Measurement
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no Liver Stiffness Measurement data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in FibroScan®/VCTE
Description: Change from baseline in Continuous Controlled Attenuation Parameter
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no Continuous Controlled Attenuation Parameter data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in FibroScan®/Vibration-controlled Transient Elastography (VCTE).
Description: Change from baseline in Fibroscan-aspartate aminotransferase (FAST) score
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no Fibroscan-aspartate aminotransferase score data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Evaluate the Effects of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Non-invasive Markers of Fibrosis and Steatosis
Description: Change from baseline in plasma pro-collagen type 3 (PRO-C3) levels
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no plasma pro-collagen type 3 data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Evaluate the Effects of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Non-invasive Markers of Fibrosis and Steatosis
Description: Change from baseline in Fibrois-4 index (FIB-4) This index is based on age, platelet count, ALT level, and AST level. FIB-4 was calculated using the following formula: FIB4 = (Age (years) x AST (U/L))/(Platelet count (10^9/L) x √ALT (U/L)).
  A decrease in FIB-4 represents a positive outcome. A FIB-4 Index of <1.45 indicates none to moderate fibrosis and an Index of >3.25 indicates advanced fibrosis.
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no Fibrois-4 index data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Evaluate the Effects of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Non-invasive Markers of Fibrosis and Steatosis
Description: Change in aspartate aminotransferase-to-platelet ratio index in Saroglitazar Magnesium groups as compared to the placebo group APRI was calculated as ([AST level/AST upper limit of normal]/ [Platelet count 1^09/L]) ×100, where AST is aspartate aminotransferase. The aspartate transaminase to platelet ratio index (APRI) is used to assess the risk of liver fibrosis.
  Higher APRI score represents a higher risk of liver fibrosis
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no aspartate aminotransferase-to-platelet ratio index data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: To Evaluate the Effects of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Non-invasive Markers of Fibrosis and Steatosis
Description: Change from baseline in Nonalcoholic fatty liver disease Fibrosis Score (NFS) The NFS is based on age, hyperglycemia, BMI, platelet count, albumin level, and AST/ALT ratio.
  NFS was calculated using the following formula: NAFLD fibrosis score = -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m^2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet (×10^9/l) - 0.66 × albumin (g/dl).
  A decrease in NFS score represents a positive outcome. An NFS score of <-1.455 indicates no advanced fibrosis and a score of >0.676 indicates liver fibrosis.
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no Nonalcoholic fatty liver disease Fibrosis Score data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Liver Enzyme
Description: Change from baseline in liver enzyme parameters (ALT and AST)
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no liver enzyme parameters (ALT and AST) data for this outcome measure were analyzed. No further data analysis for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Lipid Profile
Description: Change from baseline in triglyceride [TG), high-density lipoprotein [HDL], low-density lipoprotein [LDL], very low-density lipoprotein [VLDL], total cholesterol, and non-HDL cholesterol
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no lipid profile (triglyceride, high-density lipoprotein, low-density lipoprotein, very low-density lipoprotein, total cholesterol, non-HDL cholesterol) data for this outcome measure were analyzed. No further data analysis for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Fasting Glucose
Description: Change from baseline in fasting plasma glucose (FPG)
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no fasting plasma glucose data for this outcome measure were analyzed. No further data analysis for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Anthropometric Measurements.
Description: Change from baseline in body weight
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no body weight data for this outcome measure were analyzed. No further data analysis for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Anthropometric Measurements.
Description: Change from baseline in BMI
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no BMI data for this outcome measure were analyzed. No further data analysis for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Anthropometric Measurements.
Description: Change from baseline in hip circumference and minimum waist circumference
Time Frame: Week 24/EOT
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no hip circumference and minimum waist circumference data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: To Evaluate the Effect of Saroglitazar Magnesium 4 mg Compared With Placebo on Changes in Health-related Quality of Life Scores Measured by Short Form-36 (SF-36) Questionnaire.
Description: Change from baseline in SF-36 Questionnaire mental (MCS) and physical components scores (PCS). The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as the worst health status.
Time Frame: Week 24/EOT.
Population: The study was prematurely terminated after the enrollment of 4 participants. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. Consequently, no SF-36 Questionnaire mental (MCS) and physical components scores (PCS) data for this outcome measure were collected or analyzed. No further data collection for this specific efficacy outcome is anticipated.
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Number of Participants Experiencing Adverse Events After Consuming Saroglitazar Magnesium Compared to Placebo
Description: Number of Participants with Adverse Events. We have included data for Treatment emergent adverse events (TEAEs) only. TEAEs are those AEs that occur after administration of the study drug.
Time Frame: From baseline to Week 28
Population: The study was prematurely terminated in 29/Sep/2024 by then only 4 participants were enrolled as per V3.0 of the protocol. Due to this early termination, none of the participants reached the End of Treatment (EOT) assessment. The safety data collected was restricted to what was available up to their early discontinuation and from the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to Week 28
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saroglitazar Magnesium 4 mg (N=3) | Placebo Arm (N=1)
Upper Respiratory tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05211284/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT05211284/SAP_001.pdf